CLINICAL TRIAL: NCT01006759
Title: Proposal Evaluation and Intervention Through Prevention of Disability in Leprosy Patients
Brief Title: Prevention of Disability: Proposal for a Guidance Manual for Leprosy Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Marisa de Cássia Registro Fonseca, School of Medicine, University of Sao Paulo
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: FMRPUSP; HCRP n°14553/2005
Record Dates: First submitted 2009-11-02; First posted 2009-11-03 (Estimated); Last update posted 2009-11-03 (Estimated); Status verified 2009-11

CONDITIONS: Leprosy; Disability Evaluation; Quality of Life
Keywords: Leprosy; Disability Evaluation; Quality of Life; Sensation
MeSH Terms: conditions — Leprosy | interventions — Exercise; Counseling; Health Promotion

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- leprosy disability (Experimental): intervention of a series of cases with leprosy that made treatment in a Clinical Hospital
  Interventions: Other: exercise and orientation

INTERVENTIONS:
Other: exercise and orientation — guidances for prevention of disability in leprosy with focus on hands, eyes and feet.
  Other Names: prevention of disability; guidance; orientation; promotion of health

SUMMARY:
Leprosy is an infectious disease of slow evolution, manifested primarily by signs and symptoms dermatoneurological with skin lesions and peripheral nerve, especially in the eyes, hands and feet. The prevention of disability is essential for the control of complications. Objective: To evaluate the physical and functional status of hands, feet and eyes, for the appearance and evolution of sensory and motor deficiencies and classification of disability (WHO) of a group of leprosy patients to compare and monitor the result treatment on the progression of neuropathy and recurrence of reactions. Methodology: We performed initial physical therapy evaluation and final, after 12 months. We conducted a clinical trial of a series of 26 cases evaluated with newly diagnosed leprosy, treated by standard medication. There were used methods of qualitative and quantitative. An illustrated manual of guidelines was especially developed for this study.

DETAILED DESCRIPTION:
assessment methods of qualitative and quantitative: inspection of eyes, hands and foot, manual motor function, grip and pinch dynamometry,threshold test, SF 36 quality of life questionnaire.

Intervention: illustrated guidelines, exercises, orthoses, orientation Goals: disability prevention

ELIGIBILITY:
Inclusion Criteria:

* The patients in this project were diagnosed and referred by the dermatology to do the physical-functional evaluation and physiotherapy. We selected patients aged 18 years and both sexes, even with comorbidities, since diagnosed and treated. In accepting to participate in the research, signed a consent form

Exclusion Criteria:

* Those patients who refused to sign the consent form and those who did not attend the evaluations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2007-01; Primary Completion 2008-12 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
classification of disability for Leprosy(WHO) | 1 year

SECONDARY OUTCOMES:
classification of disability for Leprosy(WHO), grip strength and threshold sensibility | after 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Marisa CR Fonseca, PhD, Principal Investigator — University of Sao Paulo
Locations (1):
- School of Medicine, University of Sao Paulo, Ribeirão Preto, São Paulo, Brazil

REFERENCES:
- [Background] Lana FC, Amaral EP, Lanza FM, Saldanha AN. Physical disabilities resulting from Hansen's disease in Vale do Jequitinhonha/state of Minas Gerais, Brazil. Rev Lat Am Enfermagem. 2008 Nov-Dec;16(6):993-7. doi: 10.1590/s0104-11692008000600009. PMID 19229402
- See also: official website of the ministry of health — http://www.saude.gov.br